CLINICAL TRIAL: NCT04695431
Title: An External Control, Observational, Retrospective Study Assessing the Effect of Avapritinib Compared With Best Available Therapy for Patients With Advanced Systemic Mastocytosis
Brief Title: Retrospective Study Assessing the Effect of Avapritinib Versus Best Available Therapy in Patients With AdvSM
Status: Completed | Type: Observational
Sponsor: Blueprint Medicines Corporation (Industry)
Collaborators: Analysis Group, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BLU-285-2405
Record Dates: First submitted 2020-12-15; First posted 2021-01-05 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Advanced Systemic Mastocytosis; Aggressive Systemic Mastocytosis; Systemic Mastocytosis With an Associated Hematological Neoplasm; Mast Cell Leukemia
MeSH Terms: conditions — Mastocytosis, Systemic; Leukemia, Mast-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients from the BLU-285-2101 and BLU-285-2202 studies: Patients with advanced systemic mastocytosis who received treatment with avapritinib as part of the BLU-285-2101 and BLU-285-2202 studies
- External Control Group: Patients with advanced systemic mastocytosis that received best available therapy

SUMMARY:
BLU-285-2405 is a multi-center, synthetic control, observational and retrospective study designed to compare clinical outcomes for avapritinib compared with best available therapy for patients with AdvSM.

ELIGIBILITY:
Inclusion Criteria for Patients in the External Control Arm:

1. Diagnosed with AdvSM, with known subtype including SM-AHN, ASM, or MCL
2. Received at least one line of systemic therapy for AdvSM, which may include but not limited to regimens containing:

   Midostaurin Cytoreductive therapy: cladribine, interferon alpha, azacitidine, decitabine Selective TKIs: imatinib, nilotinib, dasatinib Hydroxyurea Antibody therapy: brentuximab vedotin
3. Adult (≥18 years of age) at the initiation of first systemic line of therapy at the participating site
4. Had an index date at least 3 months prior to the start of data collection (in order to include patients with at least 3 months of follow-up after index date), unless date of death occurred less than three months from index date
5. Had an approved waiver of informed consent or signed informed consent for participation in the retrospective chart review study, if no institutional waiver from the site was granted

Exclusion Criteria for Patients in the External Control Arm

1. Malignancy that is not in remission at time of SM diagnosis, or new non-hematological malignancy diagnosed after SM diagnosis, except for: completely resected basal cell and squamous cell skin cancer, curatively treated localized prostate cancer, and completely resected carcinoma in situ of any site
2. Among patients with SM-AHN, presence of either of the following:

   * Patients in whom the SM component is consistent with an indolent systemic mastocytosis (ISM) or SSM or,
   * the AHN component is a lymphoid malignancy, or one of the following myeloid malignancies: acute myeloid leukemia (AML), myelodysplastic syndrome (MDS) that is very high-or high-risk as defined by the IPSS-R, or a Philadelphia chromosome positive malignancy or,
   * there is a known FIP1L1/PDGFRA fusion gene (including those with CHIC-2 deletion and partial deletion of PDGFRA), independent of KIT mutational status
3. Received avapritinib as the first line of systemic therapy for AdvSM at participating site, or prior to initiation of first systemic therapy at participating site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients age 18 or older with a diagnosis of advanced SM.
Sampling Method: Probability Sample
Enrollment: 317 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Comparative evaluation of overall survival (OS) between patients receiving best available therapy versus avapritinib in BU-285-2101 and BLU-285-2202 | up to 12 years
  Overall Survival defined as time from initiation of systemic treatment to death from any cause

SECONDARY OUTCOMES:
Comparative evaluation between patients receiving best available therapy versus avapritinib of duration of treatment (DOT) | Up to 12 years
  DOT, defined as the duration from initiation of line of systemic treatment to discontinuation of same line of treatment for any reason and;
Comparative evaluation between patients receiving best available therapy versus avapritinib and time to next treatment line (TtNTL) | Up to 12 years
  TtNTL, defined as the time from initiation of the line of systemic treatment to the initiation of the next line of treatment
Comparative evaluation of change in serum tryptase concentration in patients receiving best available therapy versus avapritinib | Up to 12 years
  Change in serum tryptase concentration, defined as change in serum tryptase from baseline, for each line of therapy
To characterize the safety profile and conduct comparative evaluation of safety between patients receiving best available therapy vs. avapritinib | Up to 12 years
  AEs that result in treatment modification or discontinuation, hospitalization, or death according to evaluation of responsible physician

CONTACTS AND LOCATIONS:
Locations (6):
- United States (2):
  - Standford Cancer Center, Palo Alto, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
- Medizinische Universitat Wien, Vienna, Austria
- Universitatmedizin Mannheim, Mannheim, Baden-Wurttemberg, Germany
- Hospital Virgen del Valle, Toledo, Spain
- Guy's and St. Thomas' NHS Foundation Trust, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared

REFERENCES:
- [Derived] Reiter A, Gotlib J, Alvarez-Twose I, Radia DH, Lubke J, Bobbili PJ, Wang A, Norregaard C, Dimitrijevic S, Sullivan E, Louie-Gao M, Schwaab J, Galinsky IA, Perkins C, Sperr WR, Sriskandarajah P, Chin A, Sendhil SR, Duh MS, Valent P, DeAngelo DJ. Efficacy of avapritinib versus best available therapy in the treatment of advanced systemic mastocytosis. Leukemia. 2022 Aug;36(8):2108-2120. doi: 10.1038/s41375-022-01615-z. Epub 2022 Jul 5. PMID 35790816